CLINICAL TRIAL: NCT03010670
Title: Oxytocin-based Pharmacotherapy: Investigating the Effect on Interpersonal Motor Resonance Upon Direct Eye Gaze
Brief Title: Oxytocin and Interpersonal Motor Resonance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KU Leuven (Other)
Collaborators: The Branco Weiss Fellowship (Other); Research Foundation Flanders (Other)
Responsible Party: Principal Investigator, Kaat Alaerts, Prof. dr., KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: S56327b; 2014-000586-45 (EudraCT Number)
Record Dates: First submitted 2016-12-23; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2016-12

CONDITIONS: Social Behavior
Keywords: Oxytocin; Gaze processing; Interpersonal motor resonance
MeSH Terms: conditions — Social Behavior | interventions — Oxytocin; Sodium Chloride; Solutions

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin (OT) spray (Experimental): Syntocinon nasal spray (product code RVG 03716) will be used to intranasally administer one single dose (24 IU) of OT (3 puffs of 4 IU per nostril).
  Interventions: Drug: Oxytocin
- Placebo (PL) spray (Placebo Comparator): Physiological water (a solution of sodium chloride (NaCl) in water) will be used to intranasally administer one single dose (24 IU) of PL (3 puffs of 4 IU per nostril).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Oxytocin — A single dose (24IU) of nasal spray (3 puffs of 4IU per nostril) will be administered before the assessment of the neurophysiological measures.
  Other Names: Syntocinon (product code RVG 03716)
  Arms: Oxytocin (OT) spray
Other: Placebo — A single dose (24IU) of nasal spray (3 puffs of 4IU per nostril) will be administered before the assessment of the neurophysiological measures.
  Other Names: Physiological water (sodium chloride (NaCl) solution)
  Arms: Placebo (PL) spray

SUMMARY:
Among different social cues from the environment, the eyes constitute a very salient source for initiating social interaction or communication. Interestingly, previous work from our (Prinsen et al., 2016) and other labs demonstrated that direct eye contact between two individuals can readily evoke an increased propensity to 'mirror' other peoples' actions. Particularly, using transcranial magnetic stimulation (TMS), the investigators showed that mirror-motor mapping at the level of the primary motor cortex (M1), also known as "interpersonal motor resonance" (IMR), is significantly increased upon the observation of actions accompanied by direct eye contact, compared to the observation of actions accompanied by averted eye gaze.

With the present study, the investigators aim to investigate the role of eye contact on IMR further, and in particular, explore whether administration of the 'prosocial' neuropeptide oxytocin (OT) can influence eye-contact induced IMR. In general, OT is known to play an important role in promoting prosocial behavior and the perception of socially-relevant stimuli, such as eye gaze. To date however, the link between OT and IMR is less clear.

DETAILED DESCRIPTION:
In the present study, the investigators want to explore how a single-dose of intranasally administered OT can modulate interpersonal motor resonance (IMR) and/or the enhanced effects of eye contact on IMR. To investigate the effects of exogenous OT administrations, the investigators adopted a double-blind, within-subjects (cross-over), randomized, placebo-controlled trial. The investigators will recruit approximately 30 neurotypical young adults males between 18 - 35 years old. Since a cross-over design is included, subjects will participate in two sessions, separated by one week. Participants will be randomly assigned to receive a single dose of OT (24 international units) or placebo nasal spray at the first and second session.

In each session, the non-invasive brain stimulation technique 'transcranial magnetic stimulation' (TMS) will be used at the level of the primary motor cortex to obtain an end-state measure of unconscious 'mirror-motor mapping' or IMR. During TMS, participants will observe video stimuli of a model performing simple, intransitive hand movements combined with either direct or averted gaze. Additionally, behavioral measures will be included: social attachment and social responsiveness will be assessed via self-report questionnaires and eye tracking technology will be included to monitor participant's spontaneous gaze behavior.

The main statistical analysis of the neurophysiological data will have the within-subjects factor of administered nasal spray (OT or PL), observed gaze direction (direct or averted gaze) and observed movement (opening hand movement or no movement). Furthermore, the link between the neurophysiological (TMS) and behavioral measures (questionnaire data and gaze behavior) will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Young adults (between 18 - 35 y/o)
* Right-handed

Exclusion Criteria:

* Left-handed
* Any neuro(psycho)logical / psychiatric illness.
* Motor dysfunctions of the hands / arms.
* Any contradiction to TMS research as assessed with the TMS screening list: no pacemaker, implanted defibrillator, ear implant / a cochlear implant, insulin or implanted pump, a neurostimulator or ventriculoperitoneal shunt, any metallic object in the eyes (metallic fragments)

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Assessment of interpersonal motor resonance (IMR) | 30 minutes
  TMS will be applied to assess IMR during different observational conditions after a single dose of nasal spray

SECONDARY OUTCOMES:
State Adult Attachment Measure (SAAM) (sub)scores | 10 minutes
  Informant-based self-report questionnaire assessing social attachment.
Social Responsiveness Scale (SRS) (sub)scores | 20 minutes
  Informant-based self-report questionnaire assessing social responsiveness.
Spontaneous gaze behavior | 30 minutes
  During movement observation, participants' viewing behavior will be monitored by means of eye tracking technology.
Participants' mood | 10 minutes
  Informant-based self-report score on Profiles of Mood States questionnaire to control for differences in mood between sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Kaat Alaerts, PhD, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prinsen J, Bernaerts S, Wang Y, de Beukelaar TT, Cuypers K, Swinnen SP, Alaerts K. Direct eye contact enhances mirroring of others' movements: A transcranial magnetic stimulation study. Neuropsychologia. 2017 Jan 27;95:111-118. doi: 10.1016/j.neuropsychologia.2016.12.011. Epub 2016 Dec 8. PMID 27939365